CLINICAL TRIAL: NCT02562222
Title: Optimizing the Effect of Transcranial Direct Current Stimulation (tDCS) for the Treatment of Migraine
Brief Title: Optimized tDCS for the Treatment of Migraine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Optimizing_tDCS_Migraine
Record Dates: First submitted 2015-09-22; First posted 2015-09-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Migraine Disorders
Keywords: migraine disorders; transcranial direct current stimulation; electric stimulation therapy; pain; rehabilitation
MeSH Terms: conditions — Migraine Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- anodal tDCS on M1 (Experimental): anodal tDCS on left primary motor cortex
  Interventions: Procedure: anodal tDCS on M1
- cathodal tDCS on M1 (Experimental): cathodal tDCS on left primary motor cortex
  Interventions: Procedure: cathodal tDCS on M1
- anodal tDCS on V1 (Experimental): anodal tDCS on visual cortex
  Interventions: Procedure: anodal tDCS on V1
- cathodal tDCS on V1 (Experimental): cathodal tDCS on visual cortex
  Interventions: Procedure: cathodal tDCS on V1
- anodal tDCS on M1 and cathodal on V1 (Experimental): dual tDCS - anodal tDCS on left primary motor cortex and cathodal on visual cortex
  Interventions: Procedure: anodal tDCS on M1 and cathodal on V1
- cathodal tDCS on M1 and anodal on V1 (Experimental): dual tDCS - cathodal tDCS on left primary motor cortex and anodal on visual cortex
  Interventions: Procedure: cathodal tDCS on M1 and anodal on V1
- sham tDCS (Sham Comparator): sham tDCS
  Interventions: Procedure: sham tDCS

INTERVENTIONS:
Procedure: anodal tDCS on M1 — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: anodal tDCS on M1
Procedure: cathodal tDCS on M1 — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: cathodal tDCS on M1
Procedure: anodal tDCS on V1 — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: anodal tDCS on V1
Procedure: cathodal tDCS on V1 — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: cathodal tDCS on V1
Procedure: anodal tDCS on M1 and cathodal on V1 — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: anodal tDCS on M1 and cathodal on V1
Procedure: cathodal tDCS on M1 and anodal on V1 — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: cathodal tDCS on M1 and anodal on V1
Procedure: sham tDCS — The direct electric current will be applied by surface electrodes with 35cm² and composed of rubbers conductive electricity and surrounded by sponges soaked in saline solution. The electrodes position will be performed according the 10-20 international system of marking and the different montages will be realized by distinct applications sites.
  To stimuli the primary motor cortex the active electrode will be positioned on C3 point and the reference electrode on the contralateral supraorbital region. To visual cortex stimulation, the active electrode will be positioned on the Oz point and the reference on Cz. To duo stimulation, the two electrodes will be considerate actives, stimulating the visual and motor cortex simultaneously. The sham tDCS has already been used in several studies to assess the effect active tDCS and the duration of the current is only 30 seconds.
  Arms: sham tDCS

SUMMARY:
The aim of this study is to establish an optimized protocol of tDCS that normalize the lack of habituation and efficiency of inhibitory cortical circuits in migraine patients and determine tDCS polarity and the best cortical areas to stimulate which could normalize the lack of habituation and efficiency of inhibitory cortical circuits. For this, migraineurs volunteers will undergo to some tDCS protocols or sham tDCS.

DETAILED DESCRIPTION:
A crossover trial to establish an optimized tDCS protocol will be accomplished. Anodal and cathodal tDCS will be applied over the primary motor cortex (C3 - active and contralateral supra-orbital region - reference) and visual cortex (Oz - active and Cz - reference). Dual tDCS (anodal and cathodal - optimized protocol) will be applied on C3 - active and Oz - active.

Electrical cortical activity will be assessed on 14 migraineurs through: (i) MEP; (ii) MT; (iii) SICI; (iv) ICF; (v) PT and (vi) visual evoked-potential (VEP-habituation). An interval of 48hs between sessions will be taken. The order of the sessions will be randomized and counterbalanced among volunteers by site www.randomization.com.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18-55 years
* Gender: Both
* Presented diagnostic of episodic migraine with or without aura or probably migraine with or without aura according to the criteria for diagnosis of ICHD-III
* Disease duration of at least 12 months
* Without preventive medication for at least 6 months prior to initiation of treatment

Exclusion Criteria:

* Pregnant women;
* Pacemaker;
* History of seizures;
* Metallic implants in the head;
* Patients with clinical evidence of brain injuries;
* Chronic pain associated to others diseases;
* Use of neuroleptic medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Changes on VAS | through study completion, assessed up to 3 weeks (before and after each section)
  this scale will be used to measure the patients' pain intensity. VAS is an important instrument to verify, reliably, the patient's evolution during treatment. This scale will be used at beginning and end of each period (observation and treatment), before and after each tDCS session. For the VAS use, pain intensity will be asked to the patient. 0 cm means total pain absence and 10 cm is the level of maximum pain bearable by the patient.

SECONDARY OUTCOMES:
Changes on Visual Evoked Potentials measures | through study completion, assessed up to 3 weeks (before and after each section)
  volunteers will be invited to sit in a comfortable chair, in a calm and dark room, at 90 cm of distance from computer screen. It will be asked to fix his right eye visual field on a red point at the center of the screen (the left one will be blindfolded). Visual stimuli will be a black and White grid pattern, alternating at a frequency of 3.1 Hz. Electrodes used to record data will be localized on Oz and Fz points according International 10-20 system. During the test, 600 cortical answers will be recorded. Data will be collected and recorded in a personal computer, and after, converted to the ".txt" format to futures analysis with MATLAB.
Changes on motor evoked potentials | through study completion, assessed up to 3 weeks (before and after each section)
  to measure MEP, the intensity of the magnetic stimulator will be adjusted to 120% of rest motor threshold and 10 stimuli will be registered. For evaluation volunteers will be instructed to sit in a chair and get into a comfortable position. Initially, single-pulse TMS will be administered over the motor cortex to determine the cortical representation area of the first dorsal interosseous muscle (FDI). For all evaluations the same figure-eight coil is used, in order to avoid measurement bias. Amplitude means of evoked potentials will determine the MEP.
Changes on intracortical inhibition | through study completion, assessed up to 3 weeks (before and after each section)
  to evaluate these variables, subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at an inter stimulus intervals (ISI) of 2 milliseconds, to determine the short interval cortical inhibition (SICI). The Intracortical facilitation (ICF) will be evaluated by the MEP average at an ISI of 10 milliseconds. Ten stimulus will be applied in each condition (unconditioned pulse, and pairs of stimuli with ISI of 2 and 10 milliseconds). The order of stimulus delivered will be pseudorandomized and SICI and ICF will be expressed as a percentage of a conditioned stimuli in regarding an unconditioned stimuli.
Changes on intracortical facilitation | through study completion, assessed up to 3 weeks (before and after each section)
  to evaluate these variables, subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (120% of RMT) will be delivered at an inter stimulus intervals (ISI) of 2 milliseconds, to determine the short interval cortical inhibition (SICI). The Intracortical facilitation (ICF) will be evaluated by the MEP average at an ISI of 10 milliseconds. Ten stimulus will be applied in each condition (unconditioned pulse, and pairs of stimuli with ISI of 2 and 10 milliseconds). The order of stimulus delivered will be pseudorandomized and SICI and ICF will be expressed as a percentage of a conditioned stimuli in regarding an unconditioned stimuli.
Changes from phosphene threshold | through study completion, assessed up to 3 weeks (before and after each section)
  a 10-cm circular coil was used that has giving a peak magnetic field strength of 2 tesla. Subjects were asked to wear a blindfold, sit comfortably in a chair and to close their eyes to diminish ambient light.In sagittal line, three points were scored: 2, 3 and 4 cm above the inion. The single pulse TMS was applied to one of the points scored and the subject was asked to report the presence or absence of a phosphene immediately after stimulation. The stimulation was repeated ten times at each intensity with a maximum frequency of 0.2 Hz, stimulation was initially applied to 60% of the maximum intensity of the stimulator. The intensity of stimulation was changed into blocks of 5% to minimum intensity that the subject can perceive the phosphene certainly, five times ten, then this value was set as the PT.

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil